CLINICAL TRIAL: NCT00145236
Title: A Double-Blind, Multicenter, Randomized, Placebo-Controlled, Parallel Group Dosing Study of the Effects of Nebivolol on Blood Pressure in Black Patients With Mild to Moderate Hypertension.
Brief Title: Dosing Study of the Effects of Nebivolol on Blood Pressure in Black Patients With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB202
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension
Keywords: Nebivolol; Beta-Blocker
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

INTERVENTIONS:
Drug: Nebivolol

SUMMARY:
The purpose of this study was to determine if nebivolol is superior to placebo for the treatment of elevated blood pressure in Black patients with mild to moderate hypertension.

DETAILED DESCRIPTION:
This study was a Phase II, 12-week multicenter, randomized, double-blind, parallel group, placebo-controlled study of nebivolol over a range of doses in Black patients with mild to moderate hypertension. Treatment was administered once daily (qd) for 12 weeks. The study consisted of 2 phases: (1) screening/washout/single-blind placebo run-in and (2) randomization/treatment. Patients had 7 scheduled clinic visits during the study (6 clinic visits for patients not on current antihypertensive medication).

ELIGIBILITY:
Inclusion Criteria:

* Black adults with an average sitting diastolic blood pressure of greater then or equal to 95 mmHg and less then or equal to 109 mmHg at baseline.

Exclusion Criteria:

* Recent myocardial infarction or stroke
* Contraindication to beta-blocker therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-11; Study Completion 2003-08

PRIMARY OUTCOMES:
-Change in trough sitting diastolic blood pressure (DBP)at end of study compared to baseline

SECONDARY OUTCOMES:
-Change in sitting systolic blood pressure (SBP)
-Change in supine and standing DBP and SBP
-Response rate

CONTACTS AND LOCATIONS:
Overall Officials: Betty S. Riggs, MD, MBA, Study Director — Mylan Pharmaceuticals Inc
Locations (1):
- Mylan Pharmaceuticals Inc., Morgantown, West Virginia, United States